CLINICAL TRIAL: NCT07196748
Title: A Phase 3 Randomized, Double-blind, Placebo-Controlled, Parallel Group, Multicenter Protocol in Adults With an Open Label Study in Adolescents to Evaluate the Efficacy and Safety of Induction and Maintenance Therapy With Icotrokinra in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Protocol of Icotrokinra Therapy in Adult and Adolescent Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: ICONIC-UC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77242113UCO3001; 2025-521381-10-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-09-22; First posted 2025-09-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Parallel assignment applies to adult participants only.
Who Masked: Participant, Investigator
Masking Description: This study is double-blind for adults and open-label for adolescent participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Double-blind (DB) Induction Study: Icotrokinra (Experimental): Adult participants will be randomized to receive icotrokinra daily, orally starting at induction Week 0 (Week I-0). At Week I-12, all participants will be evaluated for clinical response and will enter the Maintenance study.
  Interventions: Drug: Icotrokinra
- DB Induction Study: Placebo (Placebo Comparator): Adult participants will be randomized to receive placebo daily, orally starting at Week I-0. At Week I-12, all participants will be evaluated for clinical response and will enter the Maintenance study.
  Interventions: Drug: Placebo
- DB Maintenance Study: Icotrokinra (Experimental): Adult participants who are in clinical response to icotrokinra at the end of the Induction study will enter the Maintenance study and be randomized to receive icotrokinra daily, orally starting at maintenance Week 0 (Week M-0) through Week M-40. Participants who are clinical nonresponders to icotrokinra or placebo will also enter the Maintenance study directly and receive icotrokinra daily. After completion of the Maintenance study through Week M-40, eligible participants can participate in a long-term extension (LTE).
  Interventions: Drug: Icotrokinra
- DB Maintenance Study: Placebo (Placebo Comparator): Adult participants who are in clinical response to icotrokinra at the end of the Induction study will enter the Maintenance study and be randomized to receive placebo daily, orally starting at Week M-0 through Week M-40. Participants who are clinical responders to placebo will also enter the Maintenance study directly and continue to receive placebo daily. After completion of the Maintenance study through Week M-40, eligible participants can participate in a LTE.
  Interventions: Drug: Placebo
- Open-label (OL) Induction Phase: Icotrokinra (Experimental): Adolescent participants will enter the Induction phase and receive icotrokinra daily, orally. At Week I-12 all participants will be evaluated for clinical response and will enter the Maintenance phase.
  Interventions: Drug: Icotrokinra
- OL Maintenance Phase: Icotrokinra (Experimental): Adolescent participants who are in clinical response to icotrokinra will enter the Maintenance phase at Week M-0 and continue to receive icotrokinra daily, orally up to Week M-40. Participants who are nonresponders to icotrokinra will also enter the Maintenance phase to receive icotrokinra daily. After completion of the Maintenance phase through Week M-40, eligible participants can participate in a LTE.
  Interventions: Drug: Icotrokinra

INTERVENTIONS:
Drug: Icotrokinra — Icotrokinra tablet will be administered orally.
  Other Names: JNJ-77242113
  Arms: DB Maintenance Study: Icotrokinra; Double-blind (DB) Induction Study: Icotrokinra; OL Maintenance Phase: Icotrokinra; Open-label (OL) Induction Phase: Icotrokinra
Drug: Placebo — Placebo tablet will be administered orally.
  Arms: DB Induction Study: Placebo; DB Maintenance Study: Placebo

SUMMARY:
The purpose of this protocol is to evaluate the efficacy (how well it works), safety and tolerability of oral icotrokinra as therapy in adult and adolescent participants with moderately to severely active ulcerative colitis (UC, a chronic disease of the large intestine in which the lining of the colon becomes inflamed and develops tiny open ulcers).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis (UC) established at least 12 weeks before screening including both endoscopic evidence and a histopathology report consistent with a diagnosis of UC
* Moderately to severely active UC, defined as a baseline (Week I-0) modified Mayo score of 5 to 9, inclusive, using the endoscopy subscore obtained during the central review of the screening video endoscopy
* An endoscopy subscore greater than or equal to (>=) 2 as obtained during central review of the screening video endoscopy
* For adolescent participants >=12 to less than (<) 18 years of age, body weight must be >=40 kilograms (kg) at baseline (Week I-0)
* Adult female participants of childbearing potential and all adolescent female participants must have a negative highly sensitive serum pregnancy test (beta-human chorionic gonadotropin [β-hCG]) at screening and a negative urine pregnancy test at Week I-0 prior to administration of study intervention and agree to further pregnancy tests
* Demonstrated an inadequate response, loss of response, or failure to tolerate previous conventional therapy (advanced drug therapy [ADT]-naïve) or advanced therapy defined as biologics and/or advanced oral agents for the treatment of UC (ADT-inadequate responder [IR]) as defined in the protocol

Exclusion Criteria:

* Participants with current known complications of UC such as fulminant colitis, toxic megacolon, or any other manifestation that might require colonic surgery while enrolled in the study
* Presence of a stoma
* Presence or history of a fistula
* Colonic resection within 24 weeks before baseline or any other intra-abdominal or other major surgery performed within 12 weeks before baseline
* History of extensive colonic resection (that is, less than [<] 30 centimeter [cm] of colon remaining) or colonic resection that could impair the use of disease severity assessments (for example Mayo Score) to assess response to study intervention

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 882 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-01-14 (Estimated); Study Completion 2032-01-13 (Estimated)

PRIMARY OUTCOMES:
Double-blind (DB) Induction Study: Percentage of Adult Participants in Clinical Remission at Week I-12 | At Week I-12
  Percentage of adult participants in clinical remission at Week I-12 will be reported. Clinical remission is defined as stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1.
DB Maintenance Study: Percentage of Adult Participants in Clinical Remission at Week M-40 | At Week M-40
  Percentage of adult participants in clinical remission at Week M-40 will be reported. Clinical remission is defined as stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1.
Open-Label (OL) Maintenance Phase: Percentage of Adolescent Participants in Clinical Remission at Week M-40 | At Week M-40
  Percentage of adolescent participants in clinical remission at Week M-40 will be reported. Clinical remission is defined as stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1.

SECONDARY OUTCOMES:
DB Induction Study: Percentage of Adult Participants in Clinical Response at Week I-12 | At Week I-12
  Percentage of adult participants in clinical response at Week I-12 will be reported. Clinical response is defined as a decrease from baseline in the modified Mayo score by greater than or equal to (>=) 30 percent (%) and >=2 points, with either a >=1-point decrease from baseline in the rectal bleeding subscore or a rectal bleeding subscore of 0 or 1.
DB Induction Study: Percentage of Adult Participants with Endoscopic Improvement at Week I-12 | At Week I-12
  Percentage of adult participants with endoscopic improvement at Week I-12 will be reported. Endoscopic improvement is defined as an endoscopy subscore of 0 or 1.
DB Induction Study: Percentage of Adult Participants in Symptomatic Remission at Week I-12 | At Week I-12
  Percentage of adult participants in symptomatic remission at Week I-12 will be reported. Symptomatic remission is defined as a stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0.
DB Induction Study: Percentage of Adult Participants with Inflammatory Bowel Disease Questionnaire (IBDQ) Remission at Week I-12 | At Week I-12
  Percentage of adult participants with IBDQ remission at Week I-12 will be reported. IBDQ remission is defined as an IBDQ total score of >= 170. The IBDQ is a validated, 32-item, self-reported questionnaire for participants with IBD that will be used to evaluate the disease-specific health related quality of life (HRQoL) across 4 dimensional scores: bowel symptoms (loose stools, abdominal pain), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Scores range from 32 to 224, with higher scores indicating better outcomes.
DB Induction Study: Percentage of Adult Participants with Histologic-Endoscopic Mucosal Improvement (HEMI) at Week I-12 | At Week I-12
  Percentage of adult participants with HEMI at Week I-12 will be reported. HEMI is defined as achieving a combination of histologic improvement and endoscopic improvement. Histologic improvement is defined as neutrophil infiltration in less than (<) 5% of crypts, no crypt destruction, and no erosions, ulcerations, or granulation tissue according to the Geboes grading system. Endoscopic improvement is defined as an endoscopy sub-score of 0 or 1.
DB Induction Study: Percentage of Adult Participants with Fatigue Response at Week I-12 | At Week I-12
  Percentage of adult participants with fatigue response at Week I-12 will be reported. Fatigue response is defined as a >= 7-point reduction in the patient-reported outcomes measurement information system (PROMIS)-fatigue Short Form (SF)-7a total score from baseline. The PROMIS fatigue SF-7a contains 7 items evaluating fatigue-related symptoms (that is, tiredness, exhaustion, mental tiredness, and lack of energy) and associated impacts on daily activities (that is, activity limitations related to work, self-care, and exercise).
DB Induction Study: Percentage of Adult Participants in Symptomatic Remission at Week I-4 | At Week I-4
  Percentage of adult participants in symptomatic remission at Week I-4 will be reported. Symptomatic remission is defined as a stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0.
DB Induction Study: Percentage of Adult Participants in Endoscopic Remission at Week I-12 | At Week I-12
  Percentage of adult participants in endoscopic remission at Week I-12 will be reported. Endoscopic remission is defined as an endoscopy subscore of 0.
DB Induction Study: Percentage of Adult Participants with No Bowel Urgency at Week I-12 | At Week I-12
  Percentage of adult participants with no bowel urgency at Week I-12 will be reported using the ulcerative colitis patient-reported outcomes signs and symptoms (UC-PRO/SS). The UC-PRO/SS is a 9-item measure that was developed to standardize the quantification of gastrointestinal (GI) signs and symptoms of UC through direct report from participant ratings. The module includes both bowel signs and symptoms and abdominal symptoms, with a recall period of 24 hours.
DB Induction Study: Percentage of Adult Participants with No Abdominal Pain at Week I-12 | At Week I-12
  Percentage of adult participants with no abdominal pain at Week I-12 will be reported using the UC-PRO/SS. The UC-PRO/SS is a 9-item measure that was developed to standardize the quantification of GI signs and symptoms of UC through direct report from participant ratings. The module includes both bowel signs and symptoms and abdominal symptoms, with a recall period of 24 hours.
DB Induction Study: Percentage of Adult Participants with No Bowel Incontinence at Week I-12 | At Week I-12
  Percentage of adult participants with no bowel incontinence at Week I-12 will be reported using the UC-PRO/SS. The UC-PRO/SS is a 9-item measure that was developed to standardize the quantification of GI signs and symptoms of UC through direct report from participant ratings. The module includes both bowel signs and symptoms and abdominal symptoms, with a recall period of 24 hours.
DB Induction Study: Percentage of Adult Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week I-12
  Percentage of adult participants with AEs and SAEs will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the intervention. A SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, is medically important.
DB Maintenance Study: Percentage of Adult Participants with Endoscopic Improvement at Week M-40 | At Week M-40
  Percentage of adult participants with endoscopic improvement at Week M-40 will be reported. Endoscopic improvement is defined as an endoscopy subscore of 0 or 1.
DB Maintenance Study: Percentage of Adult Participants in Symptomatic Remission at Week M-40 | At Week M-40
  Percentage of adult participants in symptomatic remission at Week M-40 will be reported. Symptomatic remission is defined as a stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0.
DB Maintenance Study: Percentage of Adult Participants with 90-day Corticosteroid-free Clinical Remission at Week M-40 | At Week M-40
  Percentage of adult participants with 90-day corticosteroid-free clinical remission at Week M-40 will be reported. 90-day corticosteroid-free clinical remission is defined as the clinical remission at the visit and not receiving corticosteroids for 90 days prior to the visit.
DB Maintenance Study: Percentage of Adult Participants with HEMI at Week M-40 | At Week M-40
  Percentage of adult participants with HEMI at Week M-40 will be reported. HEMI is defined as achieving a combination of histologic improvement and endoscopic improvement. Histologic improvement is defined as neutrophil infiltration in < 5% of crypts, no crypt destruction, and no erosions, ulcerations, or granulation tissue according to the Geboes grading system. Endoscopic improvement is defined as an endoscopy sub-score of 0 or 1.
DB Maintenance Study: Percentage of Adult Participants with IBDQ Remission at Week M-40 | At Week M-40
  Percentage of adult participants with IBDQ remission at Week M-40 will be reported. IBDQ remission is defined as an IBDQ total score of >= 170. The IBDQ is a validated, 32-item, self-reported questionnaire for participants with IBD that will be used to evaluate the disease-specific HRQoL across 4 dimensional scores: bowel symptoms (loose stools, abdominal pain), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Scores range from 32 to 224, with higher scores indicating better outcomes.
DB Maintenance Study: Percentage of Adult Participants in Endoscopic Remission at Week M-40 | At Week M-40
  Percentage of adult participants in endoscopic remission at Week M-40 will be reported. Endoscopic remission is defined as an endoscopy subscore of 0.
DB Maintenance Study: Percentage of Adult Participants in Clinical Remission at Week M-40 Among the Participants who had Achieved Clinical Remission at Maintenance Baseline | At Week M-40
  Percentage of adult participants in clinical remission at Week M-40 among the participants who had achieved clinical remission at maintenance baseline will be reported. Clinical remission is defined as stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1.
DB Maintenance Study: Percentage of Adult Participants in Histologic-Endoscopic Mucosal Remission at Week M-40 | At Week M-40
  Percentage of adult participants in histologic-endoscopic mucosal remission at Week M-40 will be reported. Histologic-endoscopic mucosal remission is defined as achieving a combination of histologic remission and endoscopic remission. Histologic remission is defined as the absence of neutrophils from the mucosa (both lamina propria and epithelium), no crypt destruction, and no erosions, ulcerations or granulation tissue according to the Geboes grading system. Endoscopic remission is defined as an endoscopy subscore of 0.
DB Maintenance Study: Percentage of Adult Participants with Fatigue Response at Week M-40 | At Week M-40
  Percentage of adult participants with fatigue response at Week M-40 will be reported. Fatigue response is defined as a >= 7-point reduction in the PROMIS-fatigue SF-7a total score from baseline. The PROMIS fatigue SF-7a contains 7 items evaluating fatigue-related symptoms (that is, tiredness, exhaustion, mental tiredness, and lack of energy) and associated impacts on daily activities (that is, activity limitations related to work, self-care, and exercise).
DB Maintenance Study: Percentage of Adult Participants with Disease Clearance at Week M-40 | At Week M-40
  Percentage of adult participants with disease clearance at Week M-40 will be reported. Disease clearance is defined as a composite of symptomatic remission and histologic-endoscopic mucosal remission. Symptomatic remission is defined as a stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0. Histologic-endoscopic mucosal remission is defined as achieving a combination of histologic remission and endoscopic remission.
DB Maintenance Study: Percentage of Adult Participants with No Bowel Urgency at Week M-40 | At Week M-40
  Percentage of adult participants with no bowel urgency at Week M-40 will be reported using the UC-PRO/SS. The UC-PRO/SS is a 9-item measure that was developed to standardize the quantification of GI signs and symptoms of UC through direct report from participant ratings. The module includes both bowel signs and symptoms and abdominal symptoms, with a recall period of 24 hours.
DB Maintenance Study: Percentage of Adult Participants with No Abdominal Pain at Week M-40 | At Week M-40
  Percentage of adult participants with no abdominal pain at Week M-40 will be reported using the UC-PRO/SS. The UC-PRO/SS is a 9-item measure that was developed to standardize the quantification of GI signs and symptoms of UC through direct report from participant ratings. The module includes both bowel signs and symptoms and abdominal symptoms, with a recall period of 24 hours.
DB Maintenance Study: Percentage of Adult Participants with No Bowel Incontinence at Week M-40 | At Week M-40
  Percentage of adult participants with no bowel incontinence at Week M-40 will be reported using the UC-PRO/SS. The UC-PRO/SS is a 9-item measure that was developed to standardize the quantification of GI signs and symptoms of UC through direct report from participant ratings. The module includes both bowel signs and symptoms and abdominal symptoms, with a recall period of 24 hours.
DB Maintenance Study: Percentage of Adult Participants with AEs and SAEs | Up to Week M-40
  Percentage of adult participants with AEs and SAEs will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the intervention. A SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, and is medically important.
OL Induction Phase: Percentage of Adolescent Participants in Clinical Response at Week I-12 | At Week I-12
  Percentage of adolescent participants in clinical response at Week I-12 will be reported. Clinical response is defined as a decrease from baseline in the modified Mayo score by greater than or equal to (>=) 30 percent (%) and >=2 points, with either a >=1-point decrease from baseline in the rectal bleeding subscore or a rectal bleeding subscore of 0 or 1.
OL Induction Phase: Percentage of Adolescent Participants in Clinical Remission at Week I-12 | At Week I-12
  Percentage of adolescent participants in clinical remission at Week I-12 will be reported. Clinical remission is defined as stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1.
OL Induction Phase: Percentage of Adolescent Participants with HEMI at Week I-12 | At Week I-12
  Percentage of adolescent participants with HEMI at Week I-12 will be reported. HEMI is defined as achieving a combination of histologic improvement and endoscopic improvement. Histologic improvement is defined as neutrophil infiltration in less than (<) 5% of crypts, no crypt destruction, and no erosions, ulcerations, or granulation tissue according to the Geboes grading system. Endoscopic improvement is defined as an endoscopy sub-score of 0 or 1.
OL Induction Phase: Percentage of Adolescent Participants with Endoscopic Improvement at Week I-12 | At Week I-12
  Percentage of adolescent participants with endoscopic improvement at Week I-12 will be reported. Endoscopic improvement is defined as an endoscopy subscore of 0 or 1.
OL Induction Phase: Percentage of Adolescent Participants in Symptomatic Remission at Week I-12 | At Week I-12
  Percentage of adolescent participants in symptomatic remission at Week I-12 will be reported. Symptomatic remission is defined as a stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0.
OL Induction Phase: Percentage of Adolescent Participants in Endoscopic Remission at Week I-12 | At Week I-12
  Percentage of adolescent participants in endoscopic remission at Week I-12 will be reported. Endoscopic remission is defined as an endoscopy subscore of 0.
OL Induction Phase: Percentage of Adolescent Participants in Pediatric Ulcerative Colitis Activity Index (PUCAI) Remission at Week I-12 | At Week I-12
  Percentage of adolescent participants in PUCAI remission at Week I-12 will be reported. PUCAI remission is defined as a PUCAI score <10. The PUCAI is a non-invasive instrument for measuring disease activity in adolescents with UC. Disease activity is determined as a score based on evaluation of abdominal pain, rectal bleeding, stool consistency, number of stools, nocturnal bowel movement, and activity level. The PUCAI score ranges from 0 to 85.
OL Induction Phase: Percentage of Adolescent Participants with AEs and SAEs | Up to Week I-12
  Percentage of adolescent participants with AEs and SAEs will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the intervention. A SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, and is medically important.
OL Maintenance Study: Percentage of Adolescent Participants with Endoscopic Improvement at Week M-40 | At Week M-40
  Percentage of adolescent participants with endoscopic improvement at Week M-40 will be reported. Endoscopic improvement is defined as an endoscopy subscore of 0 or 1.
OL Maintenance Phase: Percentage of Adolescent Participants in Symptomatic Remission at Week M-40 | At Week M-40
  Percentage of adolescent participants in symptomatic remission at Week M-40 will be reported. Symptomatic remission is defined as a stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0.
OL Maintenance Phase: Percentage of Adolescent Participants in 90-day Corticosteroid-free Clinical Remission at Week M-40 | At Week M-40
  Percentage of adolescent participants in 90-day corticosteroid-free clinical remission at Week M-40 will be reported. 90-day corticosteroid-free clinical remission is defined as the clinical remission at the visit and not receiving corticosteroids for 90 days prior to the visit.
OL Maintenance Phase: Percentage of Adolescent Participants with HEMI at Week M-40 | At Week M-40
  Percentage of adolescent participants with HEMI at Week M-40 will be reported. HEMI is defined as achieving a combination of histologic improvement and endoscopic improvement. Histologic improvement is defined as neutrophil infiltration in < 5% of crypts, no crypt destruction, and no erosions, ulcerations, or granulation tissue according to the Geboes grading system. Endoscopic improvement is defined as an endoscopy sub-score of 0 or 1.
OL Maintenance Phase: Percentage of Adolescent Participants with Histologic-Endoscopic Mucosal Remission at Week M-40 | At Week M-40
  Percentage of adolescent participants with histologic-endoscopic mucosal remission at Week M-40 will be reported. Histologic-endoscopic mucosal remission is defined as achieving a combination of histologic remission and endoscopic remission. Histologic remission is defined as the absence of neutrophils from the mucosa (both lamina propria and epithelium), no crypt destruction, and no erosions, ulcerations or granulation tissue according to the Geboes grading system. Endoscopic remission is defined as an endoscopy subscore of 0.
OL Maintenance Phase: Percentage of Adolescent Participants with Endoscopic Remission at Week M-40 | At Week M-40
  Percentage of adolescent participants with endoscopic remission at Week M-40 will be reported. Endoscopic remission is defined as an endoscopy subscore of 0.
OL Maintenance Phase: Percentage of Adolescent Participants in Clinical Remission at Week M-40 Among the Participants who had Achieved Clinical Remission at Maintenance Baseline | At Week M-40
  Percentage of adolescent participants in clinical remission at Week M-40 among the participants who had achieved clinical remission at maintenance baseline will be reported. Clinical remission is defined as stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1.
OL Maintenance Phase: Percentage of Adolescent Participants in Clinical Response at Week M-40 Among the Participants who had Achieved Clinical Response at Maintenance Baseline | At Week M-40
  Percentage of adolescent participants in clinical response at Week M-40 among the participants who had achieved clinical response at maintenance baseline will be reported. Clinical response is defined as a decrease from baseline in the modified Mayo score by >= 30 % and >=2 points, with either a >=1-point decrease from baseline in the rectal bleeding subscore or a rectal bleeding subscore of 0 or 1.
OL Maintenance Phase: Percentage of Adolescent Participants in PUCAI Remission at Week-40 | At Week M-40
  Percentage of adolescent participants in PUCAI remission at Week M-40 will be reported. PUCAI remission is defined as a PUCAI score <10. The PUCAI is a non-invasive instrument for measuring disease activity in adolescents with UC. Disease activity is determined as a score based on evaluation of abdominal pain, rectal bleeding, stool consistency, number of stools, nocturnal bowel movement, and activity level. The PUCAI score ranges from 0 to 85.
OL Maintenance Phase: Percentage of Adolescent Participants with AEs and SAEs | Up to Week M-40
  Percentage of adolescent participants with AEs and SAEs will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the intervention. A SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, and is medically important.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (193):
- United States (33):
  - AZ Gastro Care, Chandler, Arizona
  - Clinnova Research, Anaheim, California
  - Southern California Research Center, Coronado, California
  - Om Research LLC, Lancaster, California
  - TLC Clinical Research Inc, Los Angeles, California
  - GastroIntestinal Bioscience, Los Angeles, California
  - Om Research LLC, Oxnard, California
  - Clinical Applications Laboratories, Inc, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Nuvance Health Danbury Hospital, Danbury, Connecticut
  - American Institute of Research, Cutler Bay, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - GCP Clinical Research, Tampa, Florida
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - Gastroenterolgy Associates of Central GA, Macon, Georgia
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - Tri-State Gastroenterology Assoc, Crestview Hills, Kentucky
  - Delta Research Partners, LLC, West Monroe, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Westchester Putnam Gastroenterology, Carmel, New York
  - Manhattan Clinical Research LLC, New York, New York
  - New York Gastroenterology Associates, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Gastro Intestinal Research Institute of Northern Ohio LLC, Westlake, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - Susquehanna Research Group, Harrisburg, Pennsylvania
  - Digestive Disease Associates, Rock Hill, South Carolina
  - DFW Clinical Trials, Carrollton, Texas
  - Victorium Clinical Research, Houston, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
- Argentina (6):
  - GEDYT, AAI
  - Kynet Recoleta, Buenos Aires
  - CIPREC, CABA
  - Instituto de Investigaciones Clinicas T y T, Caba
  - Sanatorio Maipu, Maipú
  - HIGEA, Mendoza
- Australia (6):
  - Monash Medical Centre, Clayton
  - Concord Repatriation General Hospital, Concord
  - St Vincents Hospital Melbourne, Fitzroy
  - John Hunter Hospital, New Lambton Heights
  - Royal Melbourne Hospital, Parkville
  - Mater Hospital Brisbane, South Brisbane
- Belgium (2):
  - UZ Brussel, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
- Canada (8):
  - GIRI Gastrointestinal Research Institute, Vancouver, British Columbia
  - Viable Clinical Research, Kentville, Nova Scotia
  - Barrie GI Associates, Barrie, Ontario
  - London Digestive Disease Institute, London, Ontario
  - West GTA Research Inc, Mississauga, Ontario
  - ABP Research Services Corp., Oakville, Ontario
  - Toronto Immune and Digestive Health Institute Inc, Toronto, Ontario
  - Clinique IMD, Montreal, Quebec
- China (18):
  - China Japan Friendship Hospital, Beijing
  - Capital Medical University, Beijing Friendship Hospital, Beijing
  - Changzhou No 2 Peoples Hospital, Changzhou
  - Chongqing General Hospital, Chongqing
  - The First People's Hospital of Foshan, Foshan
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Affiliated Hospital of Hainan Medical University, Haikou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Heilongjiang Provincial Hospital, Harbin
  - Huizhou Central People's Hospital, Huizhou
  - Zhongda Hospital Southeast University, Nanjing
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - The Second Affiliatted Hospital of Soochow University, Suzhou
  - Meihekou Central Hospital, Tonghua
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuxi People s Hospital, Wuxi
  - Northern Jiangsu Peoples Hospital, Yangzhou
- Czechia (7):
  - Vojenska nemocnice Brno, Brno
  - Centrum gastroenterologie a hepatologie s.r.o., Kladno
  - PreventaMed, s.r.o., Olomouc
  - Gastromedic, Ltd., Pardubice
  - AXON Clinical s.r.o., Prague
  - Clinoxus s r o, Prague
  - MUDr. Michal Konecny, Ph.D. s.r.o., Přerov
- France (14):
  - CHU de Clermont Ferrand - Site Estaing, Clermont-Ferrand
  - APHP - Hopital Henri Mondor, Créteil
  - Institut Prive MICI Clinique des Cedres, Échirolles
  - CHU de Lille Hopital Claude Huriez, Lille
  - CHU de Limoges Hopital Dupuytren, Limoges
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - Jules Verne Clinic, Nantes
  - CHU de Nice Hopital de l Archet, Nice
  - Hopital Saint-Antoine, Paris
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - Hospices Civils de Lyon CHU Lyon Sud, Pierre-Bénite
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CHU Toulouse - Hopital de Rangueil, Toulouse
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Krankenhaus Waldfriede Mitte, Berlin
  - Medizinisches Versorgungszentrum (MVZ) Dachau, Dachau
  - Praxisgemeinschaft Jerichow, Jerichow
  - Eugastro GmbH, Leipzig
  - Universitaetsmedizin Rostock, Rostock
- Greece (2):
  - Evangelismos S A, Athens
  - University General Hospital of Heraklion, Heraklion
- Israel (11):
  - Haemek Medical Center, Afula
  - Assuta MC, Ashdod
  - Shamir Medical Center Assaf Harofeh, Be’er Ya‘aqov
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Schneider Children's Medical Center, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (32):
  - Juntendo University Hospital Urayasu, Chiba
  - Ginza central clinic, Chūōku
  - Sai Gastroenterology Proctology, Fujiidera-shi
  - Fukui Prefectural Hospital, Fukui-shi
  - Saiseikai Fukuoka General Hospital, Fukuoka
  - Gamagori City Hospital, Gamagōri
  - National Hospital Organization Mito Medical Center, Higashiibaraki-gun
  - Hirosaki General Medical Center, Hirosaki
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima
  - Kanazawa University Hospital, Kanazawa
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - Hospital of the University of Occupational and Enviromental Health, Kitakyushu
  - Kobe University Hospital, Kobe
  - Aoyama Naika Clinic, Kobe
  - Kumamoto University Hospital, Kumamoto
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Takano Hospital, Kumamoto
  - Kurume University Hospital, Kurume
  - Kyorin University Hospital, Mitaka
  - Takagi Clinic, Miyagi
  - Hyogo Medical University Hospital, Nishinomiya Shi
  - Nakagami Hospital, Okinawa
  - Kinshukai Infusion Clinic, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Japanese Red Cross Osaka Hospital, Osaka
  - Oita Red Cross Hospital, Ōita
  - Sapporo Tokushukai Hospital, Sapporo
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo
  - Matsuda Hospital, Shizuoka
  - Tokyo Metropolitan Bokutoh Hospital, Sumida Ku
  - National Hospital Organization Shizuoka Medical Center, Sunto-gun
- Malaysia (7):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Ampang, Ampang
  - Hospital Sultanah Aminah, Johor Bahru
  - Sultan Idris Shah Hospital, Kajang
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
- Poland (15):
  - Centrum Medyczne Medis ManerMed Sp Z O O, Bydgoszcz
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Vita Longa Sp z o o, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Medrise Sp. z o.o., Lublin
  - Pratia Poznan, Poznan
  - RiverMED, Poznan
  - Endoskopia Sp z o.o., Sopot
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Sonomed Sp. z o.o., Szczecin
  - GASTROMED Sp. z o.o., Torun
  - Medon Clinical Research, Warsaw
  - Bodyclinic Sp. z o.o. sp. k, Warsaw
  - Medical Network WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- Portugal (3):
  - Uls Braga - Hosp. Braga, Braga
  - Uls Loures Odivelas - Hosp. Loures, Loures
  - Ulsam - Hosp. Santa Luzia, Viana do Castelo
- Romania (2):
  - S C Delta Health Care S R L, Bucharest
  - Spitalul Clinic Colentina, Bucharest
- Spain (5):
  - Hosp. Clinic de Barcelona, Barcelona
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Virgen Macarena, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. Alvaro Cunqueiro, Vigo
- Sweden (2):
  - Ersta sjukhus, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Hospital, Ankara
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Mersin University Medical Faculty Hospital, Mersin
- United Kingdom (5):
  - Fairfield General Hospital, Greater Manchester
  - Whipps Cross University Hospital, London
  - St Georges University Hospitals NHS Foundation Trust, London
  - Whiston Hospital, Rainhill
  - Stepping Hill Hospital, Stockport

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency